CLINICAL TRIAL: NCT03853941
Title: Adherence to Activity Limitation Recommendations in Patients With Diabetic Foot Ulcers: a 'Proof of Concept' Study
Brief Title: Adherence to Activity Limitations in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 18033
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Diabetes; Foot Ulcer
Keywords: Motivation; Communication; Healthcare Professional; Training; Adherence; Diabetes; Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Communication | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in the control group will receive treatment as usual.
- Experimental (Experimental): The experimental group will receive clinical treatment as usual, however, the healthcare professionals treating them will have received training on how to enhance patient adherence via the use of a motivationally supportive communication style. Thus, the style/language healthcare professionals use to convey usual treatment recommendations may differ.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Theory-based communication training programme delivered to healthcare professionals
  Arms: Experimental

SUMMARY:
This study aims to develop and test a theory-based motivation communication training programme for healthcare professionals working with diabetic foot ulcer patients. The investigators will explore the acceptability of the training programme and examine whether the training leads to changes in healthcare professionals' communication style, and results in greater adherence to treatment recommendations (i.e., reduced weight-bearing) in patients.

DETAILED DESCRIPTION:
This is a proof of concept, two-arm non-randomised, controlled before-and-after study. Patient outcomes (perceptions of healthcare professional communication style, treatment self-regulation and adherence to activity reduction) will be collected first during a control/usual care period. Healthcare professionals will then receive the theory-based motivation communication training programme. Subsequently a new group of patients will be recruited as the intervention group and the same outcome measures collected. Control group outcomes will be compared to intervention group outcomes. Interviews will be conducted with healthcare professionals and patients to assess acceptability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 years and over
* Have diabetes according to WHO criteria
* Have a diabetic foot ulcer being treated at the foot clinic at Royal Derby Hospital
* Be able to communicate and complete questionnaire measures in English
* Have capacity to consent and agree to participate.

Exclusion Criteria:

- Patients who are not currently engaging in walking behaviour (e.g., wheelchair-bound patients) or have other physical limitations that restrict ability to use an accelerometer will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Change in healthcare professionals' communication style | Baseline
  Measured using the 6-item Health Care Climate Questionnaire, and indicated by patients' perceptions of healthcare professional autonomy support being higher in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Change in patients' adherence to activity reduction recommendations | 1 month
  Measured using an accelerometer. Patients will be asked to wear the accelerometer daily for 1 month.
Change in patient treatment self-regulation | Baseline
  Treatment self-regulation is the reasons why patients may adhere or not and is a potential mechanism explaining the relationship between healthcare professional autonomy support and patient adherence to treatment recommendations.
Acceptability of the intervention | Healthcare professional interviews 4-6 weeks following training; Patient interviews 4-6 weeks following baseline
  Assessed via interviews with healthcare professionals who have taken part in the training programme and patients.
Fidelity of delivery | Baseline
  A researcher will sit in on up to 20 patient/healthcare professional consultation sessions (10 prior to training and 10 post training). The researcher will record observations of the communication style used by the healthcare professionals within the sessions. Observations will be assessed for fidelity of delivery using a checklist developed specifically for this study. Data from pre and post-training observations will be compared for differences in communication style.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Hancox, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Royal Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No